CLINICAL TRIAL: NCT05883150
Title: Intranasal Versus Nebulized Midazolam in Behaviuor Modification of Preschool Children Undergoing Dental Treatment: A Randomized Clinical Trial
Brief Title: Intranasal Versus Nebulized Midazolam in Behaviuor Modification of Preschool Children Undergoing Dental Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 210
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dental Sedation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized Midazolam (Experimental)
  Interventions: Drug: Nebulized Midazolam
- Intranasal Midazolam (Active Comparator)
  Interventions: Drug: Intranasal Midazolam

INTERVENTIONS:
Drug: Nebulized Midazolam — All the drug solutions will be freshly prepared on the day of sedation session. Depending on the dosage calculated from the weight of each child The sedative drug, the dosage will be diluted with an equal volume by adding distilled water.
  The child will be seated in an upright position on the dental chair. Before placing the mask of the nebulizer, the child will be coached into proper breathing pattern
  Arms: Nebulized Midazolam
Drug: Intranasal Midazolam — All the drug solutions will be freshly prepared on the day of sedation session. Depending on the dosage calculated from the weight of each child, For children who will receive midazolam using the atomization device attached to a three-ml syringe, the child sitting reclined in knee-to-knee position. Half of the dose will be sprayed in the right nostril and the other half will be sprayed in the left nostril to double the absorptive surface area by short and quick puffs
  Arms: Intranasal Midazolam

SUMMARY:
The aim of the current study is to compare the effect of intranasal versus nebulized route of administration of midazolam as moderate sedative agents in preschoolers undergoing dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Frankl scale score 2.
* ASA I or II physical status.
* Dental intervention under local anesthesia not requiring more than 30 minutes.
* No previous dental experience.
* Parent/guardian's written consent.

Exclusion Criteria:

* Dental treatment indicated under general anesthesia.
* Presence of facial or nasal deformities.
* History of neurological or cognitive alterations.
* Mouth breathers

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Behavior rating | throughout the sedation session
  This will be recorded using the Modified Houpt scale for behavior rating; Sleep, head/oral resistance, crying and overall behavior will be scored on a 6-point scale ranging from 1-6 with higher scores indicating better behavior

SECONDARY OUTCOMES:
Onset of sedation | during the sedation procedure (after drug administration until reaching satisfactory sedation)
  The time taken for sedative drugs to start their action will be recorded using a stopwatch
Level of sedation | during the sedation procedure (after drug administration until reaching satisfactory sedation)
  The level of sedation Agitated will be scored using a Five point sedation scale
  * Agitated - Clinging to parent/crying
  * Alert - Awake, not clinging to parent/no cry
  * Calm - Sitting or lying comfortably with eyes spontaneously open eyes spontaneously closed but responds
  * Drowsy: Comfortable with minor stimuli
  * Asleep: Eyes closed, arousable, does not respond to minor stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Amira A ElKhatib, PhD, Principal Investigator — Kafrelsheikh University, Kafrelsheikh, Egypt; Yousr Nader, MSc, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Oral and Dental Medicine, Kafrelsheikh University, Kafrelsheikh, Egypt, Kafr ash Shaykh, Egypt